CLINICAL TRIAL: NCT02908724
Title: Cardiac Involvement in Adult Patients With Fabry Disease; Relation to Enzyme Replacement Therapy - A Nationwide Danish Clinical Cohort Study
Brief Title: Cardiac Involvement in Adult Patients With Fabry Disease; Relation to Enzyme Replacement Therapy
Status: Completed | Type: Observational
Sponsor: Ulla Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Ulla Feldt-Rasmussen, Professor, Chief physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: FAB-ECG
Record Dates: First submitted 2016-04-04; First posted 2016-09-21 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Familial cardiomyopathies; Hypertrophic cardiomyopathy; Left ventricular hypertrophy
MeSH Terms: conditions — Fabry Disease; Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ERT receiving patients: Patients that were receiving specific treatment for FD (ERT, enzyme replacement therapy, Fabrazyme or Replagal) during the observational time (n= 47).
- non-ERT receiving patients: Patients that were not receiving specific treatment for FD (ERT, enzyme replacement therapy, Fabrazyme or Replagal) during the observational time (n= 19).

SUMMARY:
The purpose of this study was to assess the progression of cardiac involvement in adult patients with Fabry Disease (FD), in the unique Danish Fabry cohort and comparing those FD patients receiving primary therapy vs. those that did not.

The hypothesis is, that we will not be able to see a significant positive difference in cardiac involvement in those FD patient who received FD specific therapy vs. those that did not.

DETAILED DESCRIPTION:
Enzyme replacement therapy and concomitant treatment:

FD specific treatment (ERT, enzyme replacement therapy) have been available since 2001 and patients have been treated with either agalsidase alpha (Replagal®) or agalsidase beta (Fabrazyme®) every other week at recommended doses, 0.2 mg/kg and 1.0 mg/kg, respectively.

Concomitant treatment with cardiovascular medication including angiotensin-converting-enzyme-inhibitor, angiotensin-II-receptor-blocker, acetylsalicylic acid, beta-blocker, calcium-channel-blocker, diuretics and statins, was registered for all patients.

Statistical analysis:

Primarily, we compared the progression of cardiac involvement from baseline to follow-up, according to ERT including subgroup analysis according to gender.

Secondarily, subgroup analysis of the ERT group was performed by separating patients with- and without cardiac disease at baseline, indicated by the presence of myocardial hypertrophy on transthoracic echocardiography (septal thickness or LV posterior wall thickness >0.9 cm for females and >1.0 for males), increased cardiac mass (Left ventricular mass index (LVMi) >95 g/m2 for females and >115g/m2 for males) or systolic dysfunction (ejection fraction <55%) in accordance with the guidelines from the American Society of Echocardiography and the European Association of Echocardiography (Lang et al., 2005).

In these analyses ERT patients' baseline was defined as the last available examination prior to ERT start and follow-up as the last available examination during ERT. Inclusion in the non-ERT group required that patient had not received ERT at study end. Intra-group comparisons of progression from baseline to follow-up were made by McNemar test (categorical variables) and Wilcoxon Signed Rank Test (continuous variables).

Thirdly, for comparisons between treatment groups, linear mixed models were applied on all available data from continuous variables regarding Sokolow-Lyon voltage-, Cornell product ECG criteria and LVMi as no violations of the assumptions for linear mixed model testing were found in initial analyses. The modelling allows for individual difference at a general level (tracking) as well as individual differences in the progression over time, controlled for gender, age at baseline, treatment duration and current ERT status.

Comparisons of major organ involvement at baseline, gene mutations and alfa-galactosidase A activity between treatment groups, were performed by Chi-squared and Mann-Whitney U tests, respectively.

Data from categorical variables are presented as frequency (percentage), and continuous variables are presented as median [range] or estimate (±standard error). Data was analysed using SPSS (version 19.0). All tests were two-sided and a p-value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Genetically verified Fabry disease
* Age at baseline >18 years
* Baseline cardiac examination performed

Exclusion Criteria:

* Switch from FD specific treatment (Fabrazyme or Replagal) to no FD specific treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty-six patients with FD
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2016-02-09 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Mass Index | Up to 13 years follow-up
  Measured by Transthoracic Echocardiography using a Philips IE 33. Two-dimensional parasternal images were used to determine left ventricular chamber dimensions and wall thickness; LV mass was calculated by the American Society of Echocardiography (ASE) equation and indexed to body surface area. Median [range] is evaluated and presented.
Left Ventricular Hypertrophy - Sokolow-Lyon voltage criteria | Up to 13 years follow-up
  12-lead electrocardiography (ECG) was performed using a Schiller Cardiovit AT-2 (Schiller AG, Dietikon, Switzerland). Left ventricular hypertrophy was evaluated by Sokolow-Lyon voltage criteria (S in V1 + R in V5/V6 ≥ 35 mm). Median [range] and frequency (%) of hypertrophy is evaluated and presented.
Left Ventricular Hypertrophy - Cornell voltage product criteria | Up to 13 years follow-up
  12-lead ECG was performed using a Schiller Cardiovit AT-2 (Schiller AG, Dietikon, Switzerland). Left ventricular hypertrophy was evaluated by Cornell product criteria (R in aVL + S in V3 (+6 mm for women) x QRS duration > 2440 mm·ms). Median [range] and frequency (%) of hypertrophy is evaluated and presented.

SECONDARY OUTCOMES:
Clinical outcome | Up to 13 years follow-up
  Cardiac interventions (medication, percutaneous coronary interventions, coronary artery bypass graft, implantation of implantable cardioverter-defibrillators or pacemakers), Cardiac symptoms (Chest pain, palpitations, edema, dyspnea, dizziness, syncope) and all-cause mortality. Frequency (%) is evaluated and presented.
Arrhythmias | Up to 13 years follow-up
  Atrial fibrillation, atrial flutter, supraventricular tachycardia, non-sustained ventricular tachycardia, measured by ECG and Holter-monitoring. Frequency (%) is evaluated and presented.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, MD,DMSc,Prof, Principal Investigator — Department of Medical Endocrinology

IPD SHARING:
Plan to Share IPD: No